CLINICAL TRIAL: NCT07337954
Title: Estimation of Critical Stone Burden Requiring JJ Stent Before Extracorporeal Shockwave Lithotripsy Using 3D-CT
Brief Title: 3D-CT vs Ellipsoid for JJ Stent Prediction Before ESWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hossam Elawady, Principal Investigator, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FMASU MS872024
Record Dates: First submitted 2025-12-26; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Urolithiasis; Shock Wave Lithotripsy; Ureteral Stents
Keywords: stone volume; 3D-CT, volumetry; stent necessity; stone burden
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Intervention Model Description: All 56 patients underwent standardized ESWL protocol (Dornier lithotripter, 2 sessions max, no initial JJ stent) with dual stone volume assessment: 3D-CT volumetry (voxel-based segmentation) vs ellipsoid formula (greatest dimensions). Patients stratified post-hoc by outcomes: success without stenting (n=14) vs complications requiring stent (n=42). No randomization; single treatment arm with diagnostic comparison
Masking Description: No masking was employed. This open-label study involved standardized ESWL treatment for all patients without initial JJ stent placement. Investigators, patients, and outcome assessors were fully aware of treatment protocol and imaging assessments (3D-CT volumetry vs ellipsoid formula). Post-hoc stratification by ESWL outcomes (success vs complications requiring stent) was performed without blinding
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESWL without Initial JJ Stent (Experimental): All 56 patients received standardized ESWL treatment using third-generation Dornier lithotripter (maximum 2 sessions, 2500 shock waves/session). No preoperative JJ stent placement. Stone volume assessed via dual methods: 3D-CT volumetry (voxel-based segmentation) and ellipsoid formula (greatest dimensions on NCCT). Follow-up at 2 weeks with KUB/ultrasound; JJ stent placed for complications (incomplete fragmentation, obstruction, Stein Strasse, infection)
  Interventions: Device: Extracorporeal shock wave lithotripter

INTERVENTIONS:
Device: Extracorporeal shock wave lithotripter — ESWL delivered at 70-80 shocks/min, max 2500 shocks/session, voltage ramped to 90 kV. Stone localization via fluoroscopy.

SUMMARY:
This prospective single-center study compares 3D-CT volumetry versus traditional ellipsoid formula to determine critical stone burden predicting JJ stent necessity before ESWL for 1-2 cm renal stones. Fifty-six patients with single radio-opaque renal stones will receive up to two ESWL sessions using Dornier lithotripter without initial stenting. Stone characteristics will be assessed via NCCT: linear dimensions (ellipsoid formula), 3D volume (voxel-based segmentation), Hounsfield units, and skin-to-stone distance. Patients will be stratified by ESWL outcomes to compare volume measurements between clearance success and stent-requiring groups..

DETAILED DESCRIPTION:
This prospective single-center study at Ain Shams University evaluates 3D-CT volumetry versus traditional ellipsoid formula for predicting critical stone burden requiring preoperative JJ stent placement in patients undergoing ESWL for 1-2 cm renal stones. Eligible patients (target n=56) with single radio-opaque renal stones will receive two ESWL sessions using Dornier lithotripter without initial stenting. Stone characteristics will be assessed via non-contrast CT (NCCT): linear dimensions (ellipsoid formula: length×width×height×0.52), 3D volume (automated voxel-based segmentation), Hounsfield units, and skin-to-stone distance.

Patients will be stratified by ESWL outcomes: stone clearance without stenting versus those requiring JJ stent due to complications (infection, incomplete fragmentation, obstruction/Stein Strasse). Volume measurements will be compared between groups using appropriate statistical tests (t-test, ROC analysis). The study aims to establish a 3D-CT volume threshold for stent prediction and validate its superiority over ellipsoid formula, particularly for irregular stone morphology.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* BMI 18-30 kg/m²
* Single radio-opaque renal stone 1-2 cm
* Suitable for ESWL per clinical assessment

Exclusion Criteria:

* Multiple renal stones
* Solitary kidney
* Impaired renal function
* Congenital renal anomalies
* Ureteric obstruction
* Systemic comorbidities
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Stone Volume by 3D-CT Volumetry | Pre-ESWL baseline
  Comparison of stone volume measured by 3D-CT volumetry (voxel-based segmentation, cm³) versus traditional ellipsoid formula (greatest dimensions method) to determine critical stone burden predicting JJ stent necessity after ESWL. ROC analysis identified optimal cutoff (>1.88 cm³) for stent requirement

SECONDARY OUTCOMES:
JJ Stent Necessity | 2 weeks post-ESWL
  Rate of JJ stent placement due to ESWL complications (incomplete fragmentation, obstruction, Stein Strasse, infection)
ESWL Success Rate | 2 weeks after maximum 2 ESWL sessions
  Stone-free rate (complete clearance or asymptomatic fragments <4mm on KUB/ultrasound)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared. Summary results are available in the publication and ClinicalTrials.gov results database.